## **Adult Caregiver Informed Consent**

**NCT number: TBD** 

Date: August 1, 2024 (last reviewed by IRB; original approval March 18, 2022)



## **Consent Form – Adult Caregiver Participation**

Dear Caregiver,

I, Dr. Kelle DeBoth Foust, Associate Professor in Occupational Therapy at Cleveland State University, am asking your permission for you to participate in a research study. For more information, please contact me at (216) 687-3628 or <a href="mailto:k.deboth@csuohio.edu">k.deboth@csuohio.edu</a>.

The purpose of this study is to understand if teaching kids and their caregivers about emotions and coping skills through a program at your child's preschool will lead to feelings of better social support, resilience, and hope. The resilience group focuses on mindfulness techniques, adaptive coping strategies, and building relationships and social supports. The focus of this resiliency training program is to provide education and introduce tools needed to overcome challenges. The intent is to improve your and/or your child's quality of life. You have been contacted about this study because the parent or legal guardian of the child you care for has identified you as a possible participant.

If you signed the consent form for your child to participate in the Resilience program, we would like to invite you to take part in a caregiver program. There is a different form to provide consent for your child. This form is for you to provide consent for yourself. The children will take part in two 8-week sessions between January and June of 2024. During that time, we will offer 3 workshops for the adult caregivers.

You will work with the occupational therapist or her assistant in a group setting with a few other caregivers for about one hour. During this time, you will engage in 3-4 structured activities, including: an icebreaker or introduction to the topic, structured activities such as adult-centered games, learning new skills, and finally a discussion of what was introduced that day. You will be asked to complete a few questionnaires for the program. These will be given to you before the program begins and after the program ends. These questionnaires should not take more than 30 minutes each time. These will assess things such as problem solving, coping skills, and stress.

This is a preliminary study. We hope the results will support use of this resiliency program for more children. I intend to present and publish the results of the study. The results will be reported as a whole. That means there is no way for anyone to identify anything about you specifically. This includes your personal scores or results. The name and specific location of the preschool will not be included publication to protect your identity.

There are minimal psychological and social risks related to participation in this study. It is also possible that you may not enjoy participating in group. Although these risks are unlikely, you will have the option not to participate should they occur. In addition, every effort will be made to be sure you feel comfortable and enjoy the group sessions. If you or the participating child are

uncomfortable or stressed at any time, you can contact the PI, Dr. Kelle DeBoth Foust. The PI will help you identify resources available to cope with stress, such as community clinics and/or social work. You can contact the PI at 216-687-3628/412-401-5143 with concerns, or by email at <a href="mailto:k.deboth@csuohio.edu">k.deboth@csuohio.edu</a>. Toll-free emotional support provided by the Ohio Department of Mental Health and Addiction Services is available 24/7 by calling their hotline at 1-800-720-9616.

There may also be a risk of confidentiality data breach, which can happen on any study. Every step will be taken to prevent this from happening. All data collected is password protected and encrypted. Any information used in future papers will not have any identifying data about you.

There are some benefits for participating. You will receive a \$25 gift card for each session that you attend. If you attend in person, small meals will be provided. You may also enjoy your time spent in group.

Reporting Child Abuse or Neglect – Ohio Revised Code

I agree to participate in the above research study.

Because the PI is a health care provider, the PI and her assistant are required to report child abuse or neglect. The Ohio Revised Code section 2151.421 requires a report to child protective services or law enforcement for cases of suspected abuse or neglect.

The alternative to participate in this study is to simply not participate. There are no costs associated with participating in this study. All needed materials will be provided to you.

Your consent and participation are voluntary. You may withdraw at any time. There is no consequence for not participating.

Please read the following: "I understand that if I have any questions about my or my child's rights as a research subject, I can contact the Cleveland State University Institutional Review Board at (216) 687-3630."

There are two copies of this form. After signing them, keep one copy for your records. Please return the other copy to your child's school. Thank you in advance for your support.

Caregiver Name: \_\_\_\_\_\_

Child's Name: \_\_\_\_\_

Caregiver's Signature: \_\_\_\_\_

Date: \_\_\_\_\_

Investigator Signature: \_\_\_\_\_